CLINICAL TRIAL: NCT00685308
Title: Wingspan Stenting for Symptomatic Severe Stenosis of Intracranial Atherosclerosis Registry in China
Acronym: WingspanSSIR
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ministry of Health, China (Other Government)
Responsible Party: Wei-Jian Jiang /Chairman of Interventional Neuroradiology, Beijing Tiantan Hospital, The Capital Medical University (CMU)
Other Study IDs: 1122837
Record Dates: First submitted 2008-05-23; First posted 2008-05-28 (Estimated); Last update posted 2008-05-28 (Estimated); Status verified 2008-05

CONDITIONS: Intracranial Atherosclerosis
Keywords: Atherosclerosis; Intracranial artery; Angioplasty; Stent
MeSH Terms: conditions — Intracranial Arteriosclerosis; Atherosclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: Stenting of atherosclerotic intracranial stenosis — Patients will receive aspirin 300mg and clopidogrel 75mg per day for 3 days or more before stenting,and for at least 1 month after stenting. Modifiable risk factors will be controlled according to major international guidelines.
  All stenting procedures will be performed in an elective setting, and under local or general anesthesia. The study will be terminated if stroke or death rate within 30 days of the stenting exceeds 15%.
  Other Names: Wingspan stenting for intracranial stenosis

SUMMARY:
This is a prospective, multi-center, non-randomized trial to study one-year outcomes of the Wingspan system for the treatment of Chinese patients with symptomatic atherosclerotic severe intracranial stenosis.

DETAILED DESCRIPTION:
The study will enroll 200 Chinese patients with atherosclerotic intracranial stenosis of 70% to 99% that causes a recent ischemic neurologic event.

The Winspan stenting following undersized Gateway balloon angioplasty will be performed at experienced centers (at least 10 cases' experiences of using the Wingspan system to treat the patients with intracranial stenosis for each center).

The primary endpoint of the study, independently evaluated by neurologists, is any stroke or death within 30 days, plus ischemic stroke in the stented artery territory between 31 day and 1 year.

ELIGIBILITY:
Inclusion Criteria:

* An angiographically verified ≥ 70% stenosis of a major intracranial artery that causes TIA or minor stroke (NIH Stroke Scale score <9) within 90 days;
* the lesion length <15 mm and normal arterial diameter adjacent to it between 2.0 mm and 4.5 mm;
* patients having at least one atherosclerotic risk factor (arterial hypertension, diabetes mellitus, hyperlipidemia, hyperhomocysteinemia and cigarette smoking).

Exclusion Criteria:

* Non-atherosclerotic stenosis;
* intracranial hemorrhage in the territory of the stenotic artery within 6 weeks; potential source of cardiac embolism;
* concurrent intracranial tumor, aneurysm and cerebral arteriovenous malformation;
* tandem >50% stenosis of extracranial carotid or vertebral artery; known contraindication to heparin, aspirin, clopidogrel, anesthesia and contrast media; hemoglobin <10 g/dl, platelet count <100,000;
* international normalized ratio >1.5 (irreversible) and uncorrectable bleeding diathesis; and life expectancy <1 years because of other medical conditions.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Chinese population with symptomatic severe stenosis of intracranial atherosclerosis
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2007-12; Primary Completion 2009-10 (Estimated); Study Completion 2010-10 (Estimated)

PRIMARY OUTCOMES:
Any stroke or death within 30 days, plus ischemic stroke in the stented artery territory between 31 day and 1 year | One year

SECONDARY OUTCOMES:
Ischemic stroke in the non-stented artery territory, hemorrhagic stroke and death from other vascular causes beyond 30 days, and emergent cerebral revascularization (ECER)and other major hemorrhages at any time within 1 year, and restenosis. | One year

CONTACTS AND LOCATIONS:
Overall Officials: Wei-Jian Jiang, MD, Principal Investigator — Beijing Tiantan Hospital, The Capital Medical University, Beijing, China
Locations (1):
- Beijiang Tiantan Hospital, The Capital Medical University, Beijing, China